CLINICAL TRIAL: NCT07176676
Title: Evaluation of the Efficacy of an Aromatherapy Treatment With Lavender Essential Oil to Reduce Post-Operative Nausea and Vomiting (PONV): Two-arm, Non-pharmacological, Single-centre, Non-profit, Randomised Controlled Trial
Brief Title: Aromatherapy Treatment With Lavender Essential Oil to Reduce Post-Operative Nausea and Vomiting (PONV)
Acronym: Leo-PONV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AziendaABCA
Record Dates: First submitted 2022-07-19; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: PONV
Keywords: nausea; vomit; lavanda; Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: Non-pharmacological, single-centre, non-profit, randomised controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender Yes (Experimental): The lavender essential oil may only be used at the first episode of nausea occurring within 24 hours post-surgery; during the same period, if nausea occurs again, it will be treated as per standard care
  Interventions: Other: Lavanda Angustifolia essential oil
- Usual Care (Active Comparator): Standard procedure, which consists of administering antiemetics if provided in therapy or reporting to the physician with a subsequent treatment decision
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Lavanda Angustifolia essential oil — Administration of Lavender Angustifolia essential oil by inhalation in reducing nausea after abdominal, vascular, neurosurgical and gynaecological surgery under general anaesthesia during the 24-hour postoperative period.
  Arms: Lavender Yes
Other: Usual Care — Patients in the Usual Care group will follow the standard procedure, which consists of administering antiemetics if provided in therapy or reporting to the doctor with a subsequent treatment decision
  Arms: Usual Care

SUMMARY:
The aim of this study is to evaluate the effectiveness of aromatherapy through the use of inhaled Lavender oil in reducing patients' nausea during the post-operative period.

DETAILED DESCRIPTION:
To evaluate the effectiveness of inhaling Lavender Angustifolia essential oil in reducing nausea after abdominal, vascular, neurosurgical and gynaecological surgery under general anaesthesia during the 24-hour postoperative period.

Secondary objective

* To detect the number of antiemetic administrations in the experimental arm compared to the control arm
* To measure the patient satisfaction of patients in the experimental group with the Lavender essential oil aromatherapy intervention at hospital discharge Primary endpoint Reduction of nausea by at least 10% compared to treatment with standard care, as assessed by the NRS (Numerical Rating Scale).

ELIGIBILITY:
Inclusion Criteria:

* Patients who sign an informed consent

  * Patients who have undergone anesthesiological examination
  * Patients undergoing general anaesthesia
  * Clinically stable patients
  * Patients with nausea scores detected with NRS>0
  * Patients admitted undergoing surgery in the Complex and/or Simple Structures listed below:
  * SC of Neurosurgery, undergoing spinal surgery
  * SC of General Surgery, undergoing surgery on one of the organs of the abdominal cavity
  * SC of Vascular Surgery, undergoing traditional surgical repair or endovascular procedure of abdominal aortic aneurysm. Sclerotherapy (to heal varicose veins) venous stripping (removal of a vein segment in the treatment of varicose veins) laser treatment
  * SS of Gynaecological Surgery, undergoing operations on the organs of the female genital apparatus.

Exclusion Criteria:

Patients with ongoing relevant cognitive impairment (Six Item Screener score <4)

* Patients with allergies or sensitivities to lavender essential oils
* Patients with asthma, COPD, Chronic Bronchitis, Obstructive Sleep Apnea
* Patients with changes in sense of smell

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of administering Lavender Angustifolia essential oil by inhalation in reducing nausea after abdominal, vascular, neurosurgical and gynaecological surgery under general anaesthesia during the 24-hour postoperative period | during the 24-hour post-operative period
  To reduce nausea after abdominal, vascular, neurosurgical and gynaecological surgery under general anaesthesia during the 24-hour postoperative period.
  Endpoint Reduction of nausea by at least 10% compared to treatment with standard care, as assessed by the NRS (Numerical Rating Scale).

SECONDARY OUTCOMES:
To evaluate the effectiveness of administering Lavender Angustifolia essential oil by inhalation in reducing nausea after abdominal, vascular, neurosurgical and gynaecological surgery under general anaesthesia during the 24-hour postoperative period | during the 24-hour postoperative period
  To measure the number of antiemetic administrations in the experimental arm compared to the control arm
o evaluate the effectiveness of administering Lavender Angustifolia essential oil by inhalation in reducing nausea after abdominal, vascular, neurosurgical and gynaecological surgery under general anaesthesia during the 24-hour postoperative period | during the 24-hour postoperative period
  To measure the patient satisfaction of the patients in the experimental group regarding the aromatherapy intervention with Lavender essential oil at hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Alessandria, Italy, Italy

IPD SHARING:
Plan to Share IPD: No